CLINICAL TRIAL: NCT03488732
Title: Valvular Heart Disease Registry - Observational Study of Percutaneous Valvular Interventions
Brief Title: Valvular Heart Disease Registry
Status: Recruiting | Type: Observational
Sponsor: Technical University of Munich (Other)
Responsible Party: Sponsor
Other Study IDs: V1
Record Dates: First submitted 2018-03-27; First posted 2018-04-05 (Actual); Last update posted 2019-04-10 (Actual); Status verified 2019-04

CONDITIONS: Valvular Heart Disease
MeSH Terms: conditions — Heart Valve Diseases | interventions — Replantation

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 10 Years
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Patients undergonig transcatheter valvular interventions
  Interventions: Device: Transcatheter valvular repair or replacement

INTERVENTIONS:
Device: Transcatheter valvular repair or replacement — Transcatheter valvular repair (predominantly MitraClip for mitral regurgitation) or replacement (predominantly transcatheter aortic valve implantation for aortic stenosis)

SUMMARY:
Patients undergoing transcatheter valvular interventions will be prospectively included into the present registry. Baseline, procedural and follow-up data will be collected and analyzed to adress various issues in the field of percutaneous valvular interventions.

ELIGIBILITY:
Inclusion Criteria:

- Severe valvular defect planned for valvular intervention

Exclusion Criteria:

- No informed consent

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Patients undergoing transcatheter valvular interventions
Sampling Method: Probability Sample
Enrollment: 2000 (Estimated)
Dates: Start 2015-04-01 (Actual); Primary Completion 2025-01-01 (Estimated); Study Completion 2030-01-01 (Estimated)

PRIMARY OUTCOMES:
All-cause mortality | 10 years

SECONDARY OUTCOMES:
Cardiovascular mortality | 10 years
NYHA status | 10 years
Grade of mitral regurgitation | 10 years

CONTACTS AND LOCATIONS:
Locations (1):
- Klinik für Innere Medizin I, München, Germany